CLINICAL TRIAL: NCT02317757
Title: Predisposing Factors Associated With Chemotherapy Toxicity in Elderly Cancer Patients: A Prospective Study
Brief Title: Predisposing Factors Associated With Chemotherapy Toxicity in Elderly Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Other Study IDs: 559/2557(EC3)
Record Dates: First submitted 2014-12-11; First posted 2014-12-16 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2016-03

CONDITIONS: Cancer
Keywords: elderly cancer patients, chemotherapy toxicity
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- cancer patients receiving chemotherapy: Patients who are older than 70 years old receiving chemotherapy

SUMMARY:
These days, there is higher proportion of elderly cancer patients. Most of them have comorbidities, borderline performance status and nutritional status. The discontinuation of chemotherapy due to unbearable toxicities was not uncommon. Comprehensive geriatric assessment might be beneficial in selection of suitable elderly patients for chemotherapy administration.

DETAILED DESCRIPTION:
The patients with the age more than 70 years old who scheduled for chemotherapy were enrolled. Geriatric assessment was performed before starting chemotherapy. The toxicity will be recorded prospectively. Predisposing factors of grade 3 and 4 toxicity will be reported.

ELIGIBILITY:
Inclusion Criteria:

* more than 70 years of age
* plan to receive first cycle of chemotherapy
* histologically or cytologically proved of cancer

Exclusion Criteria:

* patients who have concurrent chemoradiotherapy
* patients who received local chemotherapy

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: cancer patients who are older than 70 years old and receiving chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-06 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
predisposing factors of patients developed grade 3 or 4 chemotherapy toxicity | from starting chemotherapy to 1 month after last dose of chemotherapy

SECONDARY OUTCOMES:
incidence of grade 3 or 4 chemotherapy toxicity in elderly | from starting chemotherapy to 1 month after last dose of chemotherapy
Factors associated with good quality of life during receiving chemotherapy | from starting chemotherapy to 1 month after last dose of chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Suthinee Ithimakin, MD, Principal Investigator — Mahidol University
Locations (1):
- Division of medical oncology, department of medicine Siriraj Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No